CLINICAL TRIAL: NCT04372836
Title: Effect of Vasopressin Injection Technique in Laparoscopic Excision of Unilateral Ovarian Endometriomas on Ovarian Reserve: Prospective Randomized Study
Brief Title: Vasopressin Injection Technique to Preserve Ovarian Reserve in Surgery for Unilateral Ovarian Endometriomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2018-0732
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Unilateral Ovarian Endometrioma
Keywords: Endometriosis; Vasopressins; Anti-mullerian Hormone
MeSH Terms: conditions — Endometriosis; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: Primary and secondary outcomes are compared between study group and control group 6 months and 12 months after intervention during surgery for unilateral endometrioma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): During laparoscopic enucleation of unilateral endometrial cyst, no intervention is added to subjects allocated to control arm.
- Study arm (with vasopressin injection) (Experimental): During laparoscopic enucleation of unilateral endometrial cyst, diluted vasopressin is injected into the interface between endometrioma and ovarian parenchyma of patients allocated to study arm.
  Interventions: Procedure: Vasopressin injection

INTERVENTIONS:
Procedure: Vasopressin injection — The intervention consists of five steps: rupture the ovarian endometrial cyst and remove the ''chocolate fluid;'' inject diluted vasopressin solution into the interface between endometrioma and ovarian parenchyma; stop injecting until the solution overflow; separate the endometrioma away from the ovarian parenchyma; and coagulate bleeding spots and suture the ovary.
  Arms: Study arm (with vasopressin injection)

SUMMARY:
Endometriosis is a common disease with an incidence rate of 15% in women of childbearing age, and is a chronic disease that significantly affects women's quality of life by causing two problems: pain and infertility. The usual treatment for ovarian endometrioma is surgery, and the most common surgical method is laparoscopy, however, Surgery has the disadvantage of deteriorating ovarian function. Previous studies reported that local injection of vasopressin may minimize damage to the ovarian tissue during the surgical procedure. Currently, the best way to evaluate ovarian function is to measure AMH (anti-mullerian hormone). However, previous studies has not evaluated ovarian function by AMH. Aim of this study is to compare the anti-mullarian hormone (AMH) change in vasopressin-administered patients after unilateral endometrioma surgery. In this study, antimullerian hormone (AMH) will be used as an indicator of ovarian function evaluation, and will be evaluated before surgery, 6 and 12 months after surgery. Subjects were allocated randomly with stratification of AMH level 3.0mg / ml.

DETAILED DESCRIPTION:
Endometriosis is a common disease with an incidence rate of 15% in women of childbearing age, and is a chronic disease that significantly affects women's quality of life by causing two problems: pain and infertility. The usual treatment for ovarian endometrioma is surgery, and the most common surgical method is laparoscopy. Surgery has the advantage of reducing the pain of ovarian endometrioma and lower recurrence rate compared to other treatment methods, but it also has the disadvantage of deteriorating ovarian function. This is because healthy ovarian tissue adjacent to the ovarian tumor are damaged at the time of surgery, and damage to the ovarian tissue while using an electric cauterizer for hemostasis when removing the ovarian tumor. Therefore, various surgical methods have been studied to minimize damage to the ovarian tissue during the surgical procedure including local vasopressin injection into the surgical site.

Vasopressin is a peptide hormone secreted by the posterior lobe of the pituitary gland, which promotes reabsorption of water in the kidney when administered systemically, but when administered locally, it constricts blood vessels and prevents bleeding such as in esophageal variceal therapy or myomectomy. There are previous studies that demonstrated, vasopressin injection prior to endometrioma resection, the interface between the endometrioma and normal ovarian tissue is dissected, and the amount of deterioration in ovarian function after surgery is reduced compared to the group without vasopressin by reducing the amount of bleeding through vasoconstriction.

Endometriosis is the most common disease that interferes with pregnancy, and is known to have a significant decrease in ovarian function after surgery compared to other benign ovarian tumors. Currently, the best way to evaluate ovarian function is to measure AMH (anti-mullerian hormone). In a paper published in JMIG in 2014, the degradation of ovarian function was not evaluated as AMH. The purpose of this study is to investigate the effect of vasopressin on ovarian function in endometrioma surgery.

Patients who have obtained consent in advance are divided into a test group that injects vasopressin and a control that excises it without injection. In the test group, everything except the administration of vasopressin at the surgical site immediately before the endometriosis was performed is the same as that of the control group. In this study, antimullerian hormone (AMH) will be used as an indicator of ovarian function evaluation, and will be evaluated before surgery, 6 and 12 months after surgery Aim of this study is to compare the anti-mullarian hormone (AMH) change in vasopressin-administered patients after unilateral endometrioma surgery. In this study, subjects were allocated randomly with stratification of AMH level 3.0mg / ml. When α (type 1 error) = 0.05

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing laparoscopic ovarian cyst enucleation for unilateral endometrioma.
* 25≤Age≤45
* 0.5≤AMH≤7

Exclusion Criteria:

* Subjects with major medical conditions such as uncontrolled infection, diabetes, severe renal or hepatic disease.
* History of hormonal medication use within 2months

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Objective of this study is to assess decrease in ovarian reserve after ovarian endometrioma surgery.
Enrollment: 76 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
anti-mullerian hormone(AMH) | before surgery
  Anti-mullerian hormone is the most reliable marker to assess ovarian reserve to date.
anti-mullerian hormone(AMH) | 6 months after surgery
  Anti-mullerian hormone is the most reliable marker to assess ovarian reserve to date.
anti-mullerian hormone(AMH) | 12 months after surgery
  Anti-mullerian hormone is the most reliable marker to assess ovarian reserve to date.

SECONDARY OUTCOMES:
Coagulation time during surgery | during surgery
  Coagulation time has a relationship with decrease of ovarian function

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Raw data of basic dermographic informations and outcomes of interventions (AMH, coagulation time, recurrence of endometriosis cyst) can be shared.

REFERENCES:
- [Background] Saeki A, Matsumoto T, Ikuma K, Tanase Y, Inaba F, Oku H, Kuno A. The vasopressin injection technique for laparoscopic excision of ovarian endometrioma: a technique to reduce the use of coagulation. J Minim Invasive Gynecol. 2010 Mar-Apr;17(2):176-9. doi: 10.1016/j.jmig.2009.11.004. PMID 20226404
- [Background] Qiong-Zhen R, Ge Y, Deng Y, Qian ZH, Zhu WP. Effect of vasopressin injection technique in laparoscopic excision of bilateral ovarian endometriomas on ovarian reserve: prospective randomized study. J Minim Invasive Gynecol. 2014 Mar-Apr;21(2):266-71. doi: 10.1016/j.jmig.2013.07.024. Epub 2013 Sep 25. PMID 24075865
- [Background] Zhang NN, Sun TS, Yang Q. An effective "water injection"-assisted method for excision of ovarian endometrioma by laparoscopy. Fertil Steril. 2019 Sep;112(3):608-609. doi: 10.1016/j.fertnstert.2019.05.014. Epub 2019 Jul 4. PMID 31280960